CLINICAL TRIAL: NCT05154682
Title: Multi-Modal Pain Management After Outpatient Orthopaedic Surgery: A Prospective Randomized Trial
Brief Title: Pain Management After Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AILY 21D.615
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone; Tablets; Acetaminophen; Naproxen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxycodone Group (Control Group) (Active Comparator): Patients will receive oxycodone as needed after surgery
  Interventions: Drug: OxyCODONE 5 mg Oral Tablet
- Oxycodone+ Naproxen/Acetaminophen (Study Group) (Active Comparator): each patient will receive oxycodone plus acetaminophen and naproxen for 2 weeks after surgery
  Interventions: Drug: OxyCODONE 5 mg Oral Tablet; Drug: Acetaminophen 500Mg Tab; Drug: Naproxen 500 Mg

INTERVENTIONS:
Drug: OxyCODONE 5 mg Oral Tablet — Oxycodone will be given every 4 hours as needed for 2 weeks after surgery
Drug: Acetaminophen 500Mg Tab — Acetaminophen will be taken every 4 hours for 2 weeks after surgery
  Arms: Oxycodone+ Naproxen/Acetaminophen (Study Group)
Drug: Naproxen 500 Mg — Naproxen will be taken every 12 hours for 2 weeks after surgery
  Arms: Oxycodone+ Naproxen/Acetaminophen (Study Group)

SUMMARY:
Following outpatient orthopaedic surgery, adequate pain control is imperative both for patient satisfaction and for improved recovery and rehabilitation. Opioids are frequently utilized for postoperative pain control, however they can be addictive and are known to have many deleterious effects. Recent studies have demonstrated the effectiveness of a wide variety of multi-modal postoperative pain regimens in providing adequate pain control while also decreasing opioid usage. However, the most effective multi-modal pain regimen for postoperative pain control remains unclear. This prospective, randomized study intends to investigate the efficacy of a multi-modal postoperative pain regimen compared to a traditional opioid-only pain regimen following elective outpatient orthopaedic surgery of the hand, wrist, foot, or ankle.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* undergoing elective outpatient orthopaedic surgery under general anesthesia.

Exclusion Criteria:

* Age < 18 years old
* Non-English speaking
* allergy to or medical contraindication to taking oxycodone (or other opioids), acetaminophen, or Naprosyn (or other NSAIDs).
* currently taking opioid medications
* history of chronic opioid therapy for chronic pain
* surgery being performed under local anesthesia only, without general anesthesia or sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 14 days
  With the use of an 11 point numeric rating scale (NRS) daily satisfaction with their pain regimen, patients pain level and medication usage will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States